CLINICAL TRIAL: NCT00401349
Title: Immune and Inflammatory Responses in L. (Viannia) Infection Aim 2: Expression of Mif Alleles in Individuals With Recurrent Leishmaniasis, Chronic Leishmaniasis and Asymptomatic Infection
Brief Title: Expression of Mif Alleles in Individuals With Leishmaniasis
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Dr. Diane McMahon-Pratt, Yale University
Other Study IDs: 0608001742; U19AI065866 (NIH)
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2011-08

CONDITIONS: Leishmaniasis
Keywords: Leishmania; Mif Alleles; Colombia; children
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples from bucal swabs are being retained for genetic analyses of MIF alleles and possibly other genes associated with disease (leishmaniasis) resistance/susceptibility.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
CIDEIM, Centro Internacional de Entrenamiento e Investigaciones Medicas, is conducting a research study about the disease Cutaneous Leishmaniasis, which is caused by the Leishmania parasite and causes skin sores. Researchers hope to find out how the human body defends against Leishmania. A total of 472 individuals, ages 7 to 70 years, belonging to one of the following groups will be included in this study: recurring disease, chronic disease, disease with no sign or symptoms (asymptomatic), and healthy individuals. Study procedures will include a questionnaire and buccal swab (swabbing of the inside of the cheek with a cotton or wooden applicator). In addition, asymptomatic and healthy individuals will provide a blood sample. Study participation will be up to 1.5 hours.

DETAILED DESCRIPTION:
The purpose of this study is to define the proportion of low and high expression Mif alleles in individuals with recurrent or chronic Cutaneous Leishmaniasis and compare it with that of individuals with asymptomatic infection and healthy donors (controls), in order to determine if these alleles are associated with outcome of infection. This study is part 2 of a project that includes DMID protocols 05-0139 and 06-0010. Specific objectives are to: determine the proportion of low expression (5-CATT) Mif alleles in individuals with recurrent or chronic cutaneous leishmaniasis, healthy donors (controls), and individuals with asymptomatic infection; determine the proportion of high expression (6,7,8-CATT) Mif alleles in individuals with recurrent or chronic cutaneous leishmaniasis, healthy donors (controls), and individuals with asymptomatic infection; and determine the Mif Genotype repertoire and frequency distribution in the endemic population of study. This study will be conducted in 472 participants who will be enrolled into one of the following 4 groups: recurrent disease, chronic disease, asymptomatic infection, and healthy donors (controls). Patients (males and females) aged between 7-70 years with chronic or recurrent cutaneous leishmaniasis (historic or active) diagnosed in either Cali (CIDEIM) and Tumaco (San Andrés Hospital) on the Colombian Pacific Coast will be invited to participate in the study. Asymptomatic and healthy donors (controls) will also be enrolled. Pregnant women will not be enrolled. Consent and samples will be obtained during a single study visit of up to 1.5 hours. No further follow-up visits are planned for this study. Genetic material extracted and amplified from buccal swabs will be used to determine the proportion of low and high expression Mif alleles of each group. Expression in recurrent and chronic participants will be compared to that of asymptomatic participants and healthy donors (controls) in order to determine if expression frequencies are related to the outcome of infection. Blood samples obtained from asymptomatic and healthy donors will undergo in vitro blastogenesis testing to confirm asymptomatic/healthy donor status. Study outcome measures are: frequency of low expression (5-CATT) Mif alleles in participants with recurrent or chronic disease, individuals with asymptomatic infection and healthy donors (controls); frequency of high expression (6,7,8-CATT) Mif alleles in participants with recurrent or chronic disease individuals with asymptomatic infection and healthy donors (controls); and Mif Genotype repertoire and frequency distribution in the endemic population in the study site.

ELIGIBILITY:
Inclusion Criteria:

Active or historical cases of recurrent cutaneous leishmaniasis

* Age 7-70 years
* History of parasitologically confirmed (at time of diagnosis) recurrent leishmaniasis
* Voluntary participation in the study
* Written and signed Informed consent/assent forms

Active or historical cases of chronic cutaneous leishmaniasis

* Age 7-70 years
* History of parasitologically confirmed (at time of diagnosis) chronic leishmaniasis
* Voluntary participation in the study
* Written and signed Informed consent/assent forms

Asymptomatic infection

* Age 7-70 years
* Resident of endemic area
* No history or evidence of active or prior dermal leishmaniasis
* Voluntary participation in the study
* Written and signed Informed consent/assent forms

Healthy donors

* Age 7-70 years
* No history or evidence of exposure to transmission of leishmaniasis
* Voluntary participation in the study
* Written and signed Informed consent/assent forms

Exclusion Criteria:

Pregnancy

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Active or historical cases of recurrent cutaneous leishmaniasis
  2. Active or historical cases of chronic or recurrent cutaneous leishmaniasis
  3. Endemic area controls - Resident of endemic area with no history or evidence of active or prior dermal leishmaniasis
  4. Healthy donors (non-exposed to leishmaniasis)
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2006-12; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Internacional de Entrenamiento e Investigaciones Medicas, CIDEIM, Cali, Colombia